CLINICAL TRIAL: NCT05357872
Title: Dreaming During Anesthesia and Anesthetic Depth in Elective Surgery Patients Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIS and dream
Record Dates: First submitted 2021-11-25; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Dreaming; General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIS 40-50 Group (Experimental): The anesthesiologist adjusted the intravenous speed of remifentanil and propofol to maintain the bispectral index (BIS, BIS monitor; Aspect Medical System, Newton, MA) between 40-50
  Interventions: Device: deep anesthesia depth
- BIS 50-60 Group (Experimental): The anesthesiologist adjusted the intravenous speed of remifentanil and propofol to maintain the bispectral index (BIS, BIS monitor; Aspect Medical System, Newton, MA) between 50-60 during the operation.
  Interventions: Device: light anesthesia depth

INTERVENTIONS:
Device: deep anesthesia depth — The anesthesiologist adjusted the intravenous speed of remifentanil and propofol to maintain the bispectral index (BIS, BIS monitor; Aspect Medical System, Newton, MA) between 40-50 and 50-60 during the operation.
  Arms: BIS 40-50 Group
Device: light anesthesia depth — The anesthesiologist adjusted the intravenous speed of remifentanil and propofol to maintain the bispectral index (BIS, BIS monitor; Aspect Medical System, Newton, MA) between 40-50 and 50-60 during the operation.
  Arms: BIS 50-60 Group

SUMMARY:
Dreaming is a common, enduring, and fascinating part of the anesthetic experience, but its cause and timing remain elusive. Patients typically report that they were dreaming during anesthesia, but the actual timing of anesthetic dreaming is unknown. The following evidence supports the hypothesis that dreaming occurs intraoperatively and is related to light or inadequate anesthesia: (1) The incidence of dreaming has decreased as anesthetic techniques have improved; (2) dreamers exhibit more clinical signs of light anesthesia or report more awareness than non dreamers; (3) dreamers may receive lower doses of anesthetic drugs than non dreamers and emerge more rapidly from anesthesia; (4) the content of dreams may involve surgical topics or events occurring during anesthesia; and (5) in one study, the incidence of dreaming was lower in Bispectral Index (BIS)-monitored patients. Alternatively, dreaming may occur during emergence from anesthesia, when the brain is still affected by sedative concentrations of anesthetic drugs and the patient enters a sleep state. Few studies have assessed the relation between dreaming and depth of anesthesia, and their results were inconclusive.Most recently, in the B-Aware Trial, no differences in depth of anesthesia, as measured by BIS, were detected between dreamers and non dreamers. However, the patients were at high risk of awareness, and BIS data were collected manually and were only recorded in the BIS group and during maintenance. No studies investigating the relation between dreaming and depth of anesthesia during recovery were identified. Why is the investigation of dreaming during anesthesia important? Dreaming is one of the most common side effects of anesthesia but remains puzzling and requires explanation. Dreaming is sometimes distressing to patients and may decrease satisfaction with care. Some patients who report dreaming fear that their anesthetic was inadequate and that their experience was, in fact, awareness. Indeed, in a minority of cases, dreaming may truly represent near-miss awareness. The investigators therefore tested the hypothesis that dreaming during anesthesia is associated with light or inadequate anesthesia, as evidenced by higher median BIS values during maintenance of anesthesia. The investigators also explored the depth of anesthesia until emergence, the form and content of dreams, the predictors of dreaming during anesthesia, and the effect of dreaming on quality of recovery and satisfaction with anesthetic care

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years
* with an ASA physical status of I or II

Exclusion Criteria:

* presence of sleep disorders
* pain syndrome
* cardiovascular disease
* sleep apnea syndrome
* psychosis
* history of opioid usage
* history of abnormal operation or anesthesia recovery
* unwillingness to provide informed consent
* a patient with a language communication disorder

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean blood pressure | 5 minutes after entering the operation room
  record mean blood pressure during the surgery. Systolic, diastolic, or both pressures don't need to be assessed during the study period.
Mean blood pressure | procedure (anesthesia induction)
  record mean blood pressure during the surgery. Systolic, diastolic, or both pressures don't need to be assessed during the study period.
Mean blood pressure | at the end of surgery
  record mean blood pressure during the surgery. Systolic, diastolic, or both pressures don't need to be assessed during the study period.
Mean blood pressure | procedure (anesthesia extubation)
  record mean blood pressure during the surgery. Systolic, diastolic, or both pressures don't need to be assessed during the study period.
Mean blood pressure | the time when leaving the operation room
  record mean blood pressure during the surgery. Systolic, diastolic, or both pressures don't need to be assessed during the study period.
heart rate | 5 minutes after entering the operation room
  record heart rate during the surgery
heart rate | procedure (Anesthesia induction)
  record heart rate during the surgery
heart rate | at the end of surgery
  record heart rate during the surgery
heart rate | procedure (anesthesia extubation)
  record heart rate during the surgery
heart rate | the time when leaving the operation room
  record heart rate during the surgery
Bispectral Index (BIS) | 5 minutes after entering the operation room
  record BIS during the surgery. The range was 0-100. We control the range of BIS in 40-60 during the surgery
Bispectral Index (BIS) | procedure (Anesthesia induction)
  record BIS during the surgery. record BIS during the surgery. The range was 0-100. We control the range of BIS in 40-60 during the surgery
Bispectral Index (BIS) | at the end of surgery
  record BIS during the surgery. record BIS during the surgery. The range was 0-100. We control the range of BIS in 40-60 during the surgery
Bispectral Index (BIS) | procedure (anesthesia extubation)
  record BIS during the surgery. record BIS during the surgery. The range was 0-100. We control the range of BIS in 40-60 during the surgery
Bispectral Index (BIS) | the time when leaving the operation room
  record BIS during the surgery. record BIS during the surgery. The range was 0-100. We control the range of BIS in 40-60 during the surgery
Total dose of propofol | at the end of surgery
  record total dose of propofol
Dream | at the end of surgery
  Dreaming during anesthesia was defined as any experience that was described by the patient as dreaming and was thought by the patient to have occurred between the induction of anesthesia and the first moment of consciousness after anesthesia.27 Awareness was defined as postoperative recall of intraoperative events. All patients who reported dreaming were considered to be
  "dreamers" for the purpose of the analyses, whether or not they could remember the narrative of the dream. However, only dreaming reports where the narrative was remembered were classified using five-point Likert scales as follows Emotional content (1 very negative; 5 very positive) ● Memorability (1 can't remember narrative of dream; 5 most memorable ever) ● Visual vividness (1 not at all vivid; 5 most vivid ever) ● Amount of sound (1 no sound; 5 most sound ever)

SECONDARY OUTCOMES:
Postoperative adverse effects | 24 hours after surgery
  record postoperative adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: junchao zhu, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China